CLINICAL TRIAL: NCT06964529
Title: Evaluation of the Effects of I-PRF and C-PRF on Gingival Phenotype
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ümmü Gülsüm ÖĞE, Research Assistant, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024/74
Record Dates: First submitted 2025-05-01; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Gingival Phenotype; Periodontal Soft Tissue; Width of Keratinized Gingiva
Keywords: C-PRF; I-PRF; VISTA Technique

STUDY DESIGN:
Intervention Model Description: Two-arm parallel design comparing the effects of I-PRF and C-PRF on gingival phenotype using VISTA technique.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C-PRF Group (Experimental): Concentrated platelet-rich fibrin was prepared using horizontal centrifugation and injected at 4 time points (once during the VISTA procedure, and 3 additional times at 10-day intervals).
  Interventions: Biological: Concentrated PRF
- I-PRF Group (Experimental): Injectable platelet-rich fibrin was prepared using low-speed centrifugation and injected using the same protocol as C-PRF (1 surgical + 3 injection sessions).
  Interventions: Biological: Injectable PRF

INTERVENTIONS:
Biological: Concentrated PRF — Injectable platelet-rich fibrin was prepared using low-speed centrifugation and injected using the same protocol as C-PRF (1 surgical + 3 injection sessions at 10-day intervals).
  Other Names: C-PRF
  Arms: C-PRF Group
Biological: Injectable PRF — Injectable platelet-rich fibrin was prepared using low-speed centrifugation and injected using the same protocol as C-PRF (1 surgical + 3 injection sessions at 10-day intervals).
  Other Names: I-PRF
  Arms: I-PRF Group

SUMMARY:
This clinical trial aims to evaluate the effects of injectable platelet-rich fibrin (I-PRF) and concentrated platelet-rich fibrin (C-PRF) on gingival phenotype in patients undergoing mucogingival surgery with the VISTA technique. Changes in gingival thickness and width of keratinized gingiva will be assessed using both manual and digital methods.

DETAILED DESCRIPTION:
The study is designed as a randomized controlled clinical trial including 30 patients, divided into two groups: I-PRF and C-PRF. All participants receive a mucogingival procedure using the VISTA technique followed by four sessions of PRF injections (one during surgery and three at 10-day intervals). The primary outcomes are changes in gingival thickness and the width of keratinized gingiva, measured manually and digitally at baseline, 1 month, and 3 months. The aim is to compare the effectiveness of I-PRF and C-PRF on soft tissue enhancement.

ELIGIBILITY:
Inclusion Criteria:

Systemically healthy individuals aged 18-65 years No periodontal surgery in the last 6 monthsClinically healthy periodontium (no signs of active periodontal disease) Patient compliance and consent to participate

Exclusion Criteria:

Smoking Pregnancy or lactation Systemic diseases affecting healing (e.g., diabetes, immunosuppression) Use of anticoagulants or medications affecting soft tissue Poor oral hygiene or noncompliance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-08-10 (Estimated)

PRIMARY OUTCOMES:
Change in gingival thickness | Baseline, 1 month, 3 months
  Gingival thickness will be measured both manually (using a spreader) and digitally (via STL-PLY file superimposition) to assess the effect of I-PRF and C-PRF over time.

SECONDARY OUTCOMES:
Change in width of keratinized gingiva | Baseline, 1 month, 3 months
  The width of keratinized gingiva will be measured manually using a periodontal probe to evaluate the soft tissue augmentation potential of C-PRF and I-PRF.

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University Faculty of Dentistry, Malatya, Turkey (Türkiye)